CLINICAL TRIAL: NCT02784808
Title: Retrospective Analysis of Pulmonary Arterial Hypertension (PAH) and Related Complications in Juvenile Idiopathic Arthritis (JIA) Participants Treated With Biologic and Non-biologic Disease-modifying Anti-rheumatic Drugs (DMARDs)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GA29396
Record Dates: First submitted 2016-05-25; First posted 2016-05-27 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Biologic DMARDs: Participants who received biologic DMARDs as per standard of care were included in this arm.
  Interventions: Drug: Biological DMARDs
- Non-biological DMARDs: Participants who received non-biologic DMARDs as per standard of care were included in this arm.
  Interventions: Drug: Non-Biologic DMARDs

INTERVENTIONS:
Drug: Biological DMARDs — Participants will receive biologic DMARDs as per standard of CARE. The choice of specific biologic DMARD will be at the descretion of treating physician.
  Groups: Biologic DMARDs
Drug: Non-Biologic DMARDs — Participants will receive non-biologic DMARDs as per standard of care. The choice of specific non-biologic DMARD will be at the descretion of treating physician.
  Groups: Non-biological DMARDs

SUMMARY:
This study is designed to analyze the frequency and incidence rate of pulmonary complications in JIA participants who received biological DMARDs and non-biologic DMARDs. The participants having evidence of of a prescription or administration of one of the biologic or non-biologic DMARDs will be included in five different treatment groups. Data from the Thomson Reuters MarketScan® Commercial Claims and Medicare Supplemental Databases will be used to estimate the incidence rate of pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Participants with less than (<) 18 years of age at index
* Continuously enrolled for greater than (>) 6 months prior to index (baseline period)
* One diagnosis of JIA (714.3) on a non-diagnostic claim either during the baseline period (the complete participant record prior to the episode index will be defined as the episode baseline period) or within the first 30 days following the index date
* Had both medical and pharmacy benefit plus complete data availability during both baseline and follow-up periods

Exclusion Criteria:

* For biologic DMARD cohorts, prior use of any qualifying biologic belonging to the biologic DMARD of interest (using all available claims history)
* For non-biologic DMARD cohort, prior use of any non-biologic DMARD or biologic DMARD
* Any record of rituximab use in complete participant record
* A prior safety event during the baseline period

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: JIA participants treated with biologic and non-biologic DMARDs from the Thomson Reuters MarketScan® Commercial Claims and Medicare Supplemental Databases
Sampling Method: Non-Probability Sample
Enrollment: 4557 (Actual)
Dates: Start 2000-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with pulmonary arterial hypertension | up to the end of the study (up to overall period of 12 years)

SECONDARY OUTCOMES:
Percentage of participants with interstitial lung disease | up to the end of study (up to overall period of 12 years)
Percentage of participants with alveolar proteinsis | up to the end of study (approximately 2.2 years)
Percentage of participants with lipoid pneumonia | up to the end of study (up to overall period of 12 years)
Percentage of participants with pulmonary hypertension | up to the end of study (up to overall period of 12 years)
Percentage of participants with overall composite pulmonary complications | up to the end of study (up to overall period of 12 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche